CLINICAL TRIAL: NCT05170932
Title: The Use of Chlorhexidine Gel Following EDTA Root Surface Etching as an Adjunctive to Open Flap Debridement in Treating Intra-Bony Defects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2731
Record Dates: First submitted 2021-08-16; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2017-02

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Edetic Acid

STUDY DESIGN:
Intervention Model Description: chlorhexidine gel, Biological drug
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open flap + mechanical debridement (No Intervention): This group included 10 patients with periodontitis stage 2 or 3, grade A infra-bony defect sites (Caton, 2018) that had undergone proper curettage ensuring complete removal of all granulation tissue present within the defect by scaling and root planning then open flap debridement only.
- open flap +CHX gel 2 % + 24% EDTA (Experimental): This group included 10 patients with periodontitis stage 2 or 3, grade A infra-bony defect sites (Caton, 2018) that had undergone proper curettage ensuring complete removal of all granulation tissue present within the defect by scaling and root planning then open flap debridement before treating root and bony walls of the pocket surfaces by application of 24% EDTA etching and washing with saline, then application of 2% chlorhexidine gel on root surface.
  Interventions: Procedure: CHX gel 2 % + 24% EDTA

INTERVENTIONS:
Procedure: CHX gel 2 % + 24% EDTA — The local drug delivery gel (24% of EDTA gel on root and bone surface and then application of 2% of chlorhexidine gel on root surface) were placed for group 2 in the periodontal pockets Filter paper were inserted into the orifice of the pocket for 1 minute. This was done in the day of surgery then after 3 days, 7 days, 14 days and 21 days after the local drug delivery to measure the gel release profile.
  Arms: open flap +CHX gel 2 % + 24% EDTA

SUMMARY:
SUMMARY Chronic periodontitis is regarded as an inflammatory disease that affects the supporting tissues of teeth which could lead to bone destruction. According to the pattern of bone destruction, vertical infrabony defect could occur. Several biomaterials have been used to treat infrabony defects including bone grafts, membranes, anti-microbials, growth factor & Enamel matrix proteins. CHX gel which has been widely used in the treatment of infra-bony defects.

Chemical treatment of root surfaces of teeth have been used as an adjunct with mechanical instrumentation. Among these chemical agents is EDTA which was found to be able to remove the smear layer and expose the collagen fibers on the root surface which would make the root surface biocompatible favoring fibroblast attachment and increase substantivity of CHX gel. However, studies have found that there was no clinical significance of EDTA with chlorhexidine gel .

Recent studies revealed that signiﬁcant improvements could be obtained for deep intrabony defects after EDTA root surface etching and CHX gel application after non-surgical therapy compared to control non etched treated sites. This could be attributed to the associated prolonged and higher values of CHX levels for the CHX-EDTA-treated group. However, the main target of that work is to quantify levels of CHX during the early stages of healing to determine if such clinical improvement could be attributed to prolonged and increased CHX levels after EDTA root surface preconditioning.

The aim of this study was to evaluate clinically the use of Chlorhexidine gel following root surface EDTA after open flap debridement in treating Intra-bony defects and to study the effect of EDTA bone etching on Bone Morphogenetic Protein-2 (BMP-2) in gingival crevicular fluid.

DETAILED DESCRIPTION:
SUBJECTS AND METHODS A total of 20 patients were selected from the outpatient clinic of Oral Medicine, Periodontology and Oral Diagnosis department, Faculty of Dentistry, Ain Shams University. The proposal reviewed by the research ethics committee, Faculty of Dentistry, Ain-shams University.

Patients fulfilling the inclusion criteria were randomly divided into one of two groups using a randomizing program (Randomization.com):

Group 1:

This group included 10 patients with localized periodontitis stage 2 or 3, grade A infra-bony defect sites (Caton, 2018) that had undergone proper curettage ensuring complete removal of all granulation tissue present within the defect by sub-mechanical debridement then open flap debridement only.

Group 2:

This group included 10 patients with localized periodontitis stage 2 or 3, grade A infra-bony defect sites (Caton, 2018) that had undergone proper curettage ensuring complete removal of all granulation tissue present within the defect by sub-mechanical debridement then open flap debridement before treating root and bony walls of the pocket surfaces by application of 24% EDTA etching and washing with saline, then application of 2% chlorhexidine gel on root surface.

Inclusion criteria:

1. Age from 32 to 60 years old.
2. Females and males.
3. Healthy adult patients.
4. Selected patient with a single site of defect:

Two walled defect or three walled infra-bony defect. The bone defect should be at least 3 mm in depth from the crest of the alveolar bone to the base of the defect.

Pocket depth of more than or equal to 5 mm. Clinical attachment loss equal or more than 3mm.

Exclusion criteria:

1. Smokers.
2. Breast feeding and pregnant females.
3. Vulnerable group of patients (handicapped and prisoners).
4. Patients who have received any periodontal therapy or antibiotics in the last 6 months.

The study protocol explained in details to all patients. Then a signed informed consent obtained from the patients. The data obtained from patients as well as the results of the follow up will be kept confidential.

Measurements and indices:

Clinical Assessment were done using Universal Dental Williams Michigan Probe.

The following clinical parameters were measured in every patient before the surgery and after 3 months of the surgery:

Initial therapy by full mouth supra and sub-gingival mechanical debridement using ultrasonic scaler and hand instruments have been done on all patients. The patients were given instructions for self-performed plaque control measures with soft dental brush and interdental cleaning using dental floss or interdental brush to achieve good oral hygiene. All groups were subjected to the previous procedure. All groups received open flap debridement after one month of scaling and root planning.

Open flap debridement initiated by giving infiltration local anesthesia (Articaine Hydrochloride 4% and Epinephrine 1:100,000) to the affected area. Then a reverse bevel incision and full thickness flaps were elevated. This helped to gain access for deep scaling, root planning and removal of granulation tissues and tissue tags and irrigation into the pockets.

Baseline samples from the gingival crevicular fluid were collected from all selected sites using filter paper inserted into the deepest part of each periodontal pocket and left in situ for 30 seconds for assessment of BMP-2 concentrations.

In both groups, the area of selected pocket were completely dried using oil free air syringe, and then the site was isolated with cotton rolls to prevent contamination from saliva.

The local drug delivery gel (24% of EDTA gel on root and bone surface and then application of 2% of chlorhexidine gel on root surface) were placed for group 2 in the periodontal pockets using a dedicated syringe until the gel flowed out from the gingival margin for 1 minute. Filter paper were inserted into the orifice of the pocket for 1 minute. This was done in the day of surgery then after 3 days, 7 days, 14 days and 21 days after the local drug delivery to measure the gel release profile. (Ahmed Y. Gamal and Jason M. Mailhot, 2007).

The flaps were replaced as close as possible to their original position and sutured by polypropylene (4-0) suture with interrupted interproximal sutures to achieve as complete coverage of the inter-dental areas as possible.

- Poste-operative care: All patients received amoxicillin antibiotic three times per day. Patients were also prescribed 0.12% chlorhexidine digluconate mouthwash (Hexitol antiseptic mouthwash, Arab Drug Company, Egypt) to be used twice per day for one week and were instructed to avoid brushing at the site of surgery for the first ten days. Sutures were removed after 1 week and then application of perio- pack for another 1 week and follow up after 3 months.

6) Biochemical assessment: i. EDTA and Chlorhexidine gel release profile: The collected samples were labeled and carried in a dark container until High Performance Liquid Chromatography (HPLC) evaluation.

ii. Concentration of BMP-2: In both groups, assessment was done at baseline and one month after local drug delivery.

BMP-2 concentrations were determined using a commercial human BMP-2 ELISA Kit. Measurements were performed according to the manufacturer's instructions.

Measurement of BMP-2 in GCF by ELISA:

GCF was extracted from the filter paper after addition of 100ul of PBS (pH 7) and centrifugation at 5000xg. The supernatant was used for measurement of the BMP-2. The kit was provided by Chongqing Biospes Co., Ltd, China (Catalog No.: BEK1014)

ELIGIBILITY:
Inclusion criteria:

1. Age from 32 to 60 years old.
2. Females and males.
3. Healthy adult patients.
4. Selected patient with a single site of defect in single tooth:

Two walled or three walled infra-bony defect. The bone defect should be at least 3 mm in depth from the crest of the alveolar bone to the base of the defect.

Pocket depth of more than or equal to 5 mm. Clinical attachment loss equal or more than 3mm.

Exclusion criteria:

1. Smokers.
2. Breast feeding and pregnant females.
3. Vulnerable group of patients (handicapped and prisoners).
4. Patients who have received any periodontal therapy or antibiotics in the last 6 months.

The study protocol explained in details to all patients. Then a signed informed consent obtained from the patients. The data obtained from patients as well as the results of the follow up will be kept confidential.

Ages: 32 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
bleeding on probing | 3 months
  Williams graduated periodontal probe using bleeding index

SECONDARY OUTCOMES:
Bone Morphogenetic Protein-2 (BMP-2) | 3 months
  by Elissa kit release profile in gingival crevicular fluid.

OTHER OUTCOMES:
radiographic X ray | 3 months
  long parallel technique
Clinical attachment loss | 3 months
  Williams graduated periodontal probe
probing depth | 3 months
  Williams graduated periodontal probe
plaque | 3 months
  plaque index using Williams graduated periodontal probe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gamal AY, Mailhot JM. Effects of EDTA gel preconditioning of periodontally affected human root surfaces on chlorhexidine substantivity - an SEM study. J Periodontol. 2007 Sep;78(9):1759-66. doi: 10.1902/jop.2007.070124. PMID 17760546
- [Result] Gamal AY, Aziz M, Salama MH, Iacono VJ. Gingival crevicular fluid bone morphogenetic protein-2 release profile following the use of modified perforated membrane barriers in localized intrabony defects: a randomized clinical trial. J Int Acad Periodontol. 2014 Apr;16(2):55-63. PMID 24844029